CLINICAL TRIAL: NCT02055300
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Single Ascending Dose Study in Healthy Subjects to Evaluate the Safety, Tolerability and Pharmacokinetics of LY03005
Brief Title: Safety, Tolerability and Pharmacokinetics Study of LY03005
Acronym: LY03005SAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY03005
Record Dates: First submitted 2014-01-31; First posted 2014-02-05 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Meals; Desvenlafaxine Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- LY03005 - 20 (Experimental): LY03005 Dose Strength 20mg
  Interventions: Drug: LY03005; Drug: Placebo
- LY03005 - 40 (Experimental): LY03005 Dose Strength 40mg
  Interventions: Drug: LY03005; Drug: Placebo
- LY03005- 80 (Experimental): LY03005 Dose Strength 80mg
  Interventions: Drug: LY03005; Drug: Placebo
- LY03005 - 120 (Experimental): LY03005 Dose Strength 120mg
  Interventions: Drug: LY03005; Drug: Placebo
- LY03005 - 160 (Experimental): LY03005 Dose Strength 160 mg
  Interventions: Drug: LY03005; Drug: Placebo
- LY03005 - 200 (Experimental): LY03005 Dose Strength 200mg
  Interventions: Drug: LY03005; Drug: Placebo
- LY03005 - 120 - Fed (Experimental): LY03005 120mg under Fed Conditions
  Interventions: Drug: LY03005; Other: Meal
- Pristiq (Active Comparator): Pristiq - 50mg
  Interventions: Drug: Pristiq
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY03005
  Arms: LY03005 - 120; LY03005 - 120 - Fed; LY03005 - 160; LY03005 - 20; LY03005 - 200; LY03005 - 40; LY03005- 80
Drug: Placebo
  Arms: LY03005 - 120; LY03005 - 160; LY03005 - 20; LY03005 - 200; LY03005 - 40; LY03005- 80; Placebo
Other: Meal
  Arms: LY03005 - 120 - Fed
Drug: Pristiq
  Arms: Pristiq

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of escalating single oral doses of LY03005 in healthy subjects and to characterize the pharmacokinetics (PK) of escalating single oral doses of LY03005.

ELIGIBILITY:
Inclusion Criteria:

1. Are capable of giving informed consent and complying with study procedures;
2. Are between the ages of 18 and 45 years, inclusive;
3. Female subjects have a negative pregnancy test result prior to enrollment, and meet the following criteria defined as:

   1. If child-bearing potential, agree to avoid pregnancy during the study and one month after the end of the study by using at least one effective contraceptive method(s), such as an intrauterine device (IUD), diaphragm with spermicide, oral contraceptives used for at least one month prior to screening, injectable progesterone, or progesterone sub-dermal implants.
   2. Surgically sterile for at least 3 months prior to screening by one of the following means:

      * Bilateral tubal ligation
      * Salpingectomy (with or without oophorectomy)
      * Surgical hysterectomy
      * Bilateral oophorectomy (with or without hysterectomy)
   3. Postmenopausal, defined as one of the following:

      * Last menstrual period greater than 12 months prior to screening
4. Considered healthy by the Principal Investigator, based on a detailed medical history, full physical examination, clinical laboratory tests, 12-lead ECG and vital signs;
5. Nonsmoker, defined as not having smoked or used any form of tobacco in more than 6 months before screening;
6. Body mass index (BMI) of 19 to 32 kg/m2 inclusive and body weight not less than 50 kg;
7. Willing and able to adhere to study restrictions and to be confined at the clinical research center.

Exclusion Criteria:

1. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity;
2. Subjects with a mean systolic blood pressure of three measurements >130 mmHG, or a mean diastolic blood pressure of three measurements >90 mmHG at screening.
3. History or presence of malignancy other than adequately treated basal cell skin cancer
4. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody;
5. A history of seizure. However, a history of febrile seizure is allowed;
6. Positive pregnancy test result, or plan to be pregnant if female;
7. A hospital admission or major surgery within 30 days prior to screening;
8. Participation in any other investigational drug trial within 30 days from the last dosing of other trials to screening;
9. A history of prescription drug abuse, or illicit drug use within 6 months prior to screening;
10. A history of alcohol abuse according to medical history within 6 months prior to screening;
11. A positive screen for alcohol, drugs of abuse;
12. Tobacco use within 6 months prior to screening;
13. An unwillingness or inability to comply with food and beverage restrictions during study participation;
14. Donation or blood collection of more than 1 unit (approximate 450 mL) of blood (or blood products) or acute loss of blood during the 90 days prior to screening;
15. Use of prescription or over-the-counter (OTC) medications, and herbal (including St John's Wort, herbal teas, garlic extracts)within 14 days prior to dosing (Note: Use of acetaminophen at < 3g/day is permitted until 24 hours prior to dosing);
16. A history of intolerance or hypersensitivity to venlafaxine or desvenlafaxine or any excipients;
17. Patients with a history of suicide attempt in the past 6 months and/or seen by the investigator as having a significant history of risk of suicide or homicide;
18. An unwillingness of male participants to use appropriate contraceptive measures if engaging in sex intercourse with a female partner of childbearing potential. Appropriate measures include use of a condom and spermicide and, for female partners, use of an intrauterine device (IUD), diaphragm with spermicide, oral contraceptives, injectable progesterone, progesterone sub-dermal implants, or a tubal ligation. Sexual intercourse with pregnant or lactating women is prohibited.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 11 Days

SECONDARY OUTCOMES:
PK parameters of: Cmax, | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Simon Li, Study Chair — Luye Pharma Group Ltd.
Locations (1):
- Medpace, Cincinnati, Ohio, United States